CLINICAL TRIAL: NCT01774110
Title: Evaluation of Early Standardized Task-Specific Training (ESTT) in Persons With Acute Stroke
Brief Title: Evaluation of Early Standardized Task-Specific Training (ESTT)
Acronym: ESTT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very limited enrollment
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Baylor Health Care System (Other); St.David's Rehabilitation Hospital (Austin, Texas) (Unknown)
Responsible Party: Principal Investigator, Karen McCain, Associate Professor, Physical Therapy, School of Health Professions, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESTT
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Results first posted 2015-06-02 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Acute Stroke
Keywords: stroke; gait; acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- early standardized task training (Experimental): Persons in the experimental group will receive ESTT (early standardized task specific training) for gait treatment after stroke.
  Interventions: Other: Early standardized task training

INTERVENTIONS:
Other: Early standardized task training — Early standardized task training is a treatment approach using treadmill training applied very early after stroke onset.
  Other Names: ESTT

SUMMARY:
A. Specific Aims:

1. There is one specific aim of this study. The aim is to evaluate the effectiveness of early standardized task-specific training (ESTT) in persons with acute stroke.

B. Hypothesis:

1. It is our hypothesis that subjects who receive ESTT will walk faster and more symmetrically than published reports of gait outcomes in persons with stroke.

DETAILED DESCRIPTION:
It is our contention that gait recovery after stroke is impacted by the interventions that are acutely utilized during training. There is not a consensus about how to most effectively train individuals after stroke. It is clear, however, that most persons are left with significant and often debilitating gait dysfunction after stroke so there is an urgent need to find more effective therapeutic methods.

ELIGIBILITY:
Inclusion Criteria:

* Recent stroke (less than 6 weeks)
* Able to give conformed consent or have family member who can give consent
* first time stroke OR complete recovery from prior stroke

Exclusion Criteria:

* non-ambulatory before onset of stroke
* bilateral stroke
* presence of severe cardiac problems
* other co-morbidities which would affect gait training (i.e. amputation, spinal cord injury, traumatic brain injury, etc.)
* recent myocardial infarct (within 4 weeks)
* any uncontrolled health condition for which exercise is contraindicated
* severe lower extremity joint disease/pathology that would interfere with gait training
* subjects with BMI greater than 40
* significant cognitive impairment
* age greater than 80 years or less than 16 years
* able to complete 5 or more full heel raises with the affected ankle in standing with the knee extended with no more than one or two fingers on support surface for balance

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J McCain, PT, DPT, NCS, Principal Investigator — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - St. David's Rehabilitation Hospital, Austin, Texas
  - Baylor Institute for Rehabilitation - Dallas, Dallas, Texas
  - Baylor Institute for Rehabilitation - Northwest, Dallas, Texas
  - Baylor Institute for Rehabilitation - Frisco, Frisco, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Early Standardized Task Training
Started | 12
Completed | 5
Not Completed | 7
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Early Standardized Task Training
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Velocity From Initial Assessment to Completion of Study at 6 Months Post Enrollment
Description: Computerized gait analysis is done by a mat system (GAITRite) that electronically calculates the velocity.
Time Frame: This will be done at the time of discharge from inpatient rehabilitation (the initial assessment point of the study) and at 6-months post enrollment.
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | ESTT
Number analyzed (Participants) | 5
cm/sec | 35.83 (29.36)

2. Secondary Outcome: Change in Score on Stroke Rehabilitation Assessment of Movement (STREAM) Test From Initial Assessment to Discharge From Study.
Description: The Stroke Rehabilitation Assessment of Movement (STREAM) is a test of motor recovery after stroke. There are 3 subsections of the test, an upper extremity section, a lower extremity section and a mobility section. Each section is scored independently and is normed to 100 points. Each of the 3 sections is then combined into a total overall function score which is also normed to 100. Therefore, a score of 100 represents full recovery whereas a score of 50 represents about 50% recovery from the stroke.
Time Frame: This test will be done at the initiation of the protocol (initial assessment) and at 6 months post enrollment
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Early Standardized Treadmill Training
Number analyzed (Participants) | 5
scores on a scale | 28.63 (13.78)

3. Other Pre Specified Outcome: Change in 6-Minute Walk Test Distance From Time of Discharge From Rehabilitation (Initial Assessment) to 6 Months Post Enrollment
Description: The 6-Minute Walk Test is a test of walking endurance and walking velocity.
Time Frame: This test will be done at the initiation of the protocol (initial assessment) and at 6 months post enrollment
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Early Standardized Treadmill Training
Number analyzed (Participants) | 5
feet | 448.66 (215.77)

ADVERSE EVENTS:
Time Frame: 1.5 years
Description: no adverse events were reported
Groups:
- ESTT: early standardized treadmill training
Arm/Group | ESTT
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No